CLINICAL TRIAL: NCT04979832
Title: A Combined Treatment With GM-CSF, Fosfomycin and Metronidazole for Pouchitis in Ulcerative Colitis Patients After Restorative Ileal Pouch Anal Anastomosis Surgery
Brief Title: GM-CSF, Fosfomycin and Metronidazole for Pouchitis in Ulcerative Colitis Patients After Restorative IPAA Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REG-106-2020; 2020-000609-10 (EudraCT Number)
Record Dates: First submitted 2021-06-30; First posted 2021-07-28 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Pouchitis
MeSH Terms: conditions — Pouchitis | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Fosfomycin; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Local administration of GM-CSF, fosfomycin and metronidazole in the pouch (Experimental): Local administration of 50 micrograms GM-CSF, 400 milligrams fosfomycin and 100 milligrams metronidazole in the pouch.
  In a Phase A of the trial, this will be applied as a single dose during endoscopy of the pouch. In Phase B of the trial, this will be applied as a first dose during endoscopy of the pouch, followed by 6 further daily doses for a total of 7 doses.
  Interventions: Drug: GM-CSF, fosfomycin and metronidazole

INTERVENTIONS:
Drug: GM-CSF, fosfomycin and metronidazole — GM-CSF 50 micrograms Fosfomycin 400 milligrams Metronidazole 100 milligrams applied as a gel in the pouch
  Other Names: GM-CSF; Fosfomycin; Metronidazole

SUMMARY:
This study will examine whether the application of GM-CSF, fosfomycin and metronidazole locally in the pouch is safe and effective in the treatment of pouchitis for patients with ulcerative colitis, and whether treatment changes the microbiome of the pouch.

DETAILED DESCRIPTION:
A definitive cure for patients with treatment-refractory ulcerative colitis is proctocolectomy with IPAA (restorative ileal pouch anal anastomosis). Up to 50% of all patients develop "pouchitis" within the first five years after surgery, an inflammatory condition that is as yet poorly understood and without official consensus on treatment. Treatment modalities include oral antibiotics as well as immunomodulators, steroids, probiotics and biological agents, but up to 20% of these patients develop chronic, treatment-resistant pouchitis, which can result in pouch failure and the need for reoperation with the possible creation of an ileostomy.

The etiology of pouchitis is thought to be similar to other inflammatory bowel diseases, in that genetic and bacterial factors, a compromised gastrointestinal barrier and immunological components seem to play a role. Its pathogenetic mechanisms seem to mimic Crohn's disease, in which smaller studies have shown some effect of systemically administered GM-CSF (granulocyte-macrophage colony stimulating factor) on the gut macrophage function in clearing microorganisms and maintaining the mucosal barrier.

The investigators hypothesize that GM-CSF will have an effect in the treatment of pouchitis because of its similarity to that of Crohn's disease. In order to maximize effect on the inflamed mucosa and minimize systemic side effects, the study drug will be administered locally in the pouch. In a safety and proof-of-concept intervention study, 50 µg GM-CSF will be combined with 400 mg Fosfomycin and 100 mg Metronidazole, to target both the suspected immunological as well as the bacterial role in the pathogenesis of pouchitis.

The effect on the pouch will be assessed endoscopically and histologically by taking biopsies that will also be examined for changes in the microbiome. Trial participants will be clinically examined and have blood samples taken to monitor for adverse reactions. The primary outcome measure will be an assessment of adverse reactions and tolerability of the drug. Secondary outcome measures will be a change in the pouchitis disease activity index (PDAI), a change in the microbial diversity, and a change in inflammatory markers.

This study is based on a non-randomized trial design with an open-label single group assignment.

Phase I The tolerability of treatment will be tested on 6 trial participants with pouchitis with a single dose of the combined medication applied endoscopically in the pouch. Endoscopy with the taking of biopsies will be performed before and one week after administration of the medication, as well as blood samples before and after the medication. After the follow-up endoscopy, the trial participant will receive standard oral metronidazole or ciprofloxacin treatment for 10 days.

Phase II Depending on effect of the first study, the second study plans for the treatment of 12 trial participants. Endoscopy with biopsies will be conducted with the first application of the study drug combination in the pouch, and afterward a daily dosage for another 6 days. Clinical and endoscopic control after 14 days with blood samples and biopsies will be done. After the follow-up endoscopy, the trial participant will receive standard oral metronidazole or ciprofloxacin treatment for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Of any gender
* Over 18 years of age
* Have a previous diagnosis of ulcerative colitis
* Have had IPAA surgery, and
* Have been diagnosed with pouchitis
* Be able to understand and complete study procedures as determined by the investigator
* Be able to speak either Danish or English
* Be able to comply with study procedures for the length of the study
* Use a highly effective contraception method for the duration of the trial (until day 30 in Phase I and until day 37 in Phase II), such as implants, injectables, oral contraceptives, IUD (intrauterine device), sexual abstinence or vasectomized partner.

Exclusion Criteria:

* Patients with a previous allergic reaction to GM-CSF, metronidazole or fosfomycin
* Patients who are currently under antibiotic treatment or have received antibiotic treatment within the past 30 days
* Patients currently pregnant or breastfeeding
* Patients with ASA IV classification (American Society of Anesthesiologists physical status classification)
* Patients with severe pulmonary disease
* Patients with autoimmune thrombocytopenia
* Patients with severe renal impairment (eGFR < 40 ml/min)
* Patients with alcohol use disorder or history of drug abuse
* Patients currently in treatment for any malignant or hematological disease
* Patients with a previous history of cancer will be excluded from the study (except for patients with well-treated and stabile cancer after a control period of more than two years).
* Patients with anticipated compliance problems as determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1: safety study, Determine serious adverse reactions or adverse reactions from the application of GM-CSF, metronidazole and fosfomycin in the pouch | 30 days after first application of study drug
  Incidence of Treatment-Emergent Adverse Events
Phase 2: Proof of concept study, Change in the pouchitis disease activity index (PDAI) | 14 days after first application of the study drug
  A decrease of 3 points or more will be determined as an improvement in PDAI from before application of the study drug to 7 days after application of the study drug. Between 0-18 points can be given, with a score of 7 or higher indicating pouchitis.

SECONDARY OUTCOMES:
Phase 1: Change in the pouchitis disease activity index (PDAI) | Within 7 days after application of the study drug
  A decrease of 3 points or more will be determined as an improvement in PDAI from before application of the study drug to 7 days after application of the study drug. Between 0-18 points can be given, with a score of 7 or higher indicating pouchitis.
Phase 1: Number of trial participants with a change in median white blood cells after treatment | Within 7 days after application of the study drug
  Change in median white blood cells (numbers × 10^9/L)
Phase 1: Number of trial participants with a change in median CRP after treatment | Within 7 days after application of the study drug
  Change in median CRP (mg/L)
Phase 1: Number of trial participants with a change in median creatinine after treatment | Within 7 days after application of the study drug
  Change in median creatinine (µmol/L)
Phase 1: Number of trial participants with a change in median liver enzymes after treatment | Within 7 days after application of the study drug
  Change in median liver enzymes (ALAT, alanine-aminotransferase in U/L)
Phase 1: Change in microbial diversity in the pouch using 16S rRNA sequencing | Within 7 days after application of the study drug
  A qualitative assessment of the microbial diversity of the mucosa of the pouch by determining species names and distribution quantity using 16S rRNA sequencing.
Phase 2: Change in the clinical, endoscopic or histological PDAI | 14 days after first application of the study drug
  A decrease of 3 points or more will be determined as an improvement in PDAI individually for clinical (0-6 points), endoscopic (0-6 points) and histological (0-6 points) PDAI.
Phase 2: Number of trial participants with a change in median white blood cells after treatment | 14 days after first application of the study drug
  Change in median white blood cells (numbers × 10^9/L)
Phase 2: Number of trial participants with a change in median CRP after treatment | 14 days after first application of the study drug
  Change in median CRP (mg/L)
Phase 2: Number of trial participants with a change in median creatinine after treatment | 14 days after first application of the study drug
  Change in median creatinine (µmol/L)
Phase 2: Number of trial participants with a change in median liver enzymes after treatment | 14 days after first application of the study drug
  Change in median liver enzymes (ALAT, alanine-aminotransferase in U/L)
Phase 2: Change in microbial diversity in the pouch using 16S rRNA sequencing | 14 days after first application of the study drug
  A qualitative assessment of the microbial diversity of the mucosa of the pouch by determining species names and distribution quantity using 16S rRNA sequencing.
Phase 2: Determine serious adverse reactions or adverse reactions from the application of GM-CSF, metronidazole and fosfomycin in the pouch | 37 days after first application of the study drug
  Incidence of Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Gögenur, Professor, Principal Investigator — Zealand University Hospital
Locations (1):
- Zealand University Hospital, Køge, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT04979832/Prot_000.pdf
  • Informed Consent Form (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT04979832/ICF_001.pdf